**Official Title:** The Effect of Dental Anxiety on the Success of Mandibular Anesthesia in Mandibular Molar Teeth with Symptomatic Irreversible Pulpitis: A Prospective Clinical Study

NCT Number: Not available

**Date:** 15/12/2024

Null Hypothesis (H<sub>0</sub>): Dental anxiety does not affect the success of mandibular anesthesia in the treatment of symptomatic irreversible pulpitis in mandibular molar teeth.

**Study arms:** A prospective clinical trial with two parallel intervention arms. Participants will be divided into two groups based on their Modified Dental Anxiety Scale (MDAS) scores:

- Group 1 (Low Anxiety Group): MDAS score < 10
- Group 2 (Moderate to High Anxiety Group): MDAS score ≥ 11 (including those with dental phobia if MDAS > 19)

Sample Size Calculation: Using G\*Power 3.1.9.7 software, based on an effect size of 0.8,  $\alpha = 0.05$ , and power = 0.80, the required sample size was determined as **26 patients per group**, totaling **52 participants**. The actual power achieved was 81%.

## **Materials and Methods:**

## **Inclusion Criteria:**

- o Systemically healthy adults aged 18–65
- Mandibular molar teeth with symptomatic irreversible pulpitis requiring root canal treatment
- o Radiographic evidence of closed apex and absence of periapical pathology
- o Periodontal probing depth  $\leq 3 \text{ mm}$
- o Tooth mobility < 0.5 mm
- Pain score of 55–170 mm on the Heft-Parker Visual Analog Scale (HP-VAS) (i.e., moderate or severe pain)

0

## • Exclusion Criteria:

- Systemic disease
- o Teeth with open apex, periapical lesion, internal or external resorption
- Periodontal probing depth > 3 mm
- $\circ$  Tooth mobility > 0.5 mm
- o HP-VAS score < 55 mm (no or mild pain)
- Pregnant patients or those with allergy to articaine

#### **Procedure:**

- All treatments and measurements will be conducted between 09:00 and 12:00 to minimize circadian and cortisol fluctuations.
- Patients will avoid food intake for at least 2 hours before treatment and abstain from caffeine, alcohol, tobacco, and intense exercise within 24 hours.
- Patients will rest in the dental chair for 5 minutes, then their demographic data will be recorded.
- MDAS will be administered to assess anxiety level.
- HP-VAS will be used to assess pre-treatment pain level.
- Pulse rate, SpO<sub>2</sub>, and salivary cortisol levels will be recorded pre- and post-anesthesia.

#### **Anesthesia Protocol:**

- All procedures are performed by a single operator in a one-unit room.
- Topical anesthesia: 10% lidocaine spray (Locanest) applied for 60 seconds.
- IANB (Inferior Alveolar Nerve Block):
  - 1.8 ml of 4% articaine hydrochloride with 1:100,000 epinephrine (Ultracaine DS Forte)
    via 27G needle
- Buccal and lingual infiltration:
  - o Additional 1.8 ml injection performed 5 minutes after IANB
- Block Failure Definition:
  - o If deep lip numbness is not achieved within 15 minutes, the block is considered failed and the participant is withdrawn from the study.

# **Outcome Evaluation:**

- During treatment, if the patient feels pain, they raise their hand, and the pain is marked on the HP-VAS.
- If required, supplemental anesthesia (PDL or intrapulpal) will be administered and recorded.
- Successful anesthesia: No or mild discomfort
- Failed anesthesia: Moderate or severe pain
- Cold test will be performed 15 minutes after IANB. If positive, additional anesthesia will be given.

# **Biological Sampling:**

- Saliva samples will be collected 15 minutes before and after anesthesia.
- Samples will be stored at -80°C until analysis.
- Special sterile, single-use Sali-Tubes (SLV-4158, DRG, Germany) will be used.

# **Statistical Analysis:**

All statistical analyses will be performed using SPSS Statistics 20 software (IBM Corp., Armonk, NY) at a 5% significance level. If the data are normally distributed, Student's t-test will be used to compare preoperative pain levels, salivary cortisol, SpO<sub>2</sub>, and pulse rate across different anxiety levels. Chisquare test will be used to analyze the relationship between anxiety levels and the success rate of anesthesia.